CLINICAL TRIAL: NCT07003373
Title: Comparison of the Pregnancy Outcomes of Frozen Embryo Transfer in the Natural Cycle vs. Artificial Cycle
Brief Title: Comparison of Two Protocols in Frozen Embryo Transfer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malihe Mahmoudinia (Other)
Responsible Party: Sponsor-Investigator, Malihe Mahmoudinia, Associate Professor of obstetrics & Gynecology, Fellowship of infertility, Faculty of Medicine, Mashhad University of Medical Sciences, Mashhad, Iran, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.MUMS.IRH.REC.1403.221
Record Dates: First submitted 2025-04-25; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: IVF Outcomes
Keywords: Natural cycle; Artificial cycle; Frozen embryo transfer
MeSH Terms: interventions — Hormone Replacement Therapy; Population Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural cycle group (No Intervention): A transvaginal ultrasound is performed on cycle day 2 or 3 to rule out ovarian cysts and confirm an endometrial thickness <5 mm. If eligible, patients are monitored from day 8 onward. Ovulation is tracked by assessing dominant follicle growth (≥15 mm), LH surge (≥17 IU/L), and serum progesterone (>1.5 ng/mL). Once ovulation is confirmed and endometrial thickness reaches ≥7 mm, FET is scheduled for 6 days post-LH surge or 5 days post-follicle collapse. Serum progesterone is measured one day before transfer; if <10 ng/mL, 400 mg/day progesterone is administered
- Hormone Replacement Therapy (HRT) (Experimental)
  Interventions: Drug: hormone replacement therapy (HRT) group

INTERVENTIONS:
Drug: hormone replacement therapy (HRT) group — Estradiol valerate is initiated at 4 mg/day on day 2 of the menstrual cycle and is adjusted to 8 mg/day based on endometrial thickness. Once the endometrial thickness reaches ≥8 mm, progesterone supplementation is started (400 mg vaginal suppositories twice daily and 50 mg intramuscular injections daily) for 5 days before blastocyst transfer.
  Arms: Hormone Replacement Therapy (HRT)

SUMMARY:
This randomized clinical trial evaluates two different endometrial preparation protocols-hormone replacement therapy (HRT) and natural cycle-for frozen embryo transfer (FET) in infertile women undergoing assisted reproductive technology (ART). The goal is to compare implantation, clinical pregnancy, and ongoing pregnancy outcomes.

DETAILED DESCRIPTION:
This prospective, randomized controlled clinical trial is conducted on women aged 18 to 42 years undergoing frozen embryo transfer (FET) during in vitro fertilization (IVF) cycles. Eligible participants meet the inclusion criteria and provide written informed consent.

Participants are randomized into two groups using a permuted block method:

HRT Group (Control): Estradiol valerate is initiated at 4 mg/day on day 2 of the menstrual cycle and is adjusted to 8 mg/day based on endometrial thickness. Once the endometrial thickness reaches ≥8 mm, progesterone supplementation is started (400 mg vaginal suppositories twice daily and 50 mg intramuscular injections daily) for 5 days before blastocyst transfer.

Natural Cycle Group: A transvaginal ultrasound is performed on cycle day 2 or 3 to rule out ovarian cysts and confirm an endometrial thickness <5 mm. If eligible, patients are monitored from day 8 onward. Ovulation is tracked by assessing dominant follicle growth (≥15 mm), LH surge (≥17 IU/L), and serum progesterone (>1.5 ng/mL). Once ovulation is confirmed and endometrial thickness reaches ≥7 mm, FET is scheduled for 6 days post-LH surge or 5 days post-follicle collapse. Serum progesterone is measured one day before transfer; if <10 ng/mL, 400 mg/day progesterone is administered.

Embryos are cultured in Blastocyst medium (Origio, Denmark) and assessed daily. High-quality embryos (Grade A) are defined by a 4-cell stage on day 2, a 7-8 cell stage on day 3, uniform cell size, and <20% fragmentation. Blastocyst grading follows Gardner's criteria. One or two top-quality embryos are transferred using a Cook catheter under abdominal ultrasound guidance. If no blastocyst is available by day 5, the most advanced embryo is transferred.

ELIGIBILITY:
Inclusion Criteria:

Regular menstrual cycles

Maternal age between 18 and 42 years

Normal intrauterine cavity confirmed by pretreatment ultrasound or hysteroscopy

Body Mass Index (BMI) less than 30 kg/m²

No ovulation disorders

Exclusion Criteria:

No embryos available for transfer (no embryo thawing)

Withdrawal of patient consent to continue treatment

Failure of dominant follicle development (in natural cycle group)

Inadequate endometrial response for transfer

No endometriosis grade 3 or higher

The participant provided written informed consent

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks post-transfer
  presence of gestational sac on ultrasound at 6 weeks
Chemical pregnancy rate | 12-16 days post embryo transfer
  Positive BHCG test greater than 25 mIU/ml after 12-16 days of embryo transfer

SECONDARY OUTCOMES:
Ongoing Pregnancy Rate | At 20 weeks after embryo transfer
  Pregnancy sustained beyond 20 weeks gestation
Early Miscarriage Rate | Up to 12 weeks after embryo transfer
  loss of a fetus before 12 weeks of gestation
Late Miscarriage Rate | up to 24 weeks gestation
  loss of a fetus after 12 weeks and before 24 weeks
Live Birth Rate | At delivery, After 24 weeks gestation
  Birth of at least one live neonate after 24 completed weeks of gestation
Cycle Cancellation Rate | Up to the day of embryo transfer
  Proportion of treatment cycles canceled before embryo transfer
Pregnancy Complications | through study completion, an average of 1 year
  Incidence of pregnancy-related complications, including: Preeclampsia: Onset of hypertension after 20 weeks of gestation, Gestational Diabetes, Placental Abruption,Placenta Previa

IPD SHARING:
Plan to Share IPD: Undecided